CLINICAL TRIAL: NCT07290673
Title: A Multicenter, Prospective, Randomized Controlled Trial Evaluating the Efficacy of Foundation DRS Solo as an Adjunct to Standard of Care Versus Standard of Care Alone in the Treatment of Nonhealing Diabetic Foot Ulcers.
Brief Title: Evaluating the Efficacy of FoundationDRS Solo in Addition to Standard of Care for the Treatment of Non-healing Diabetic Foot Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samaritan Biologics (Industry)
Collaborators: Emergent Clinical Consulting, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SB-25-1
Record Dates: First submitted 2025-10-30; First posted 2025-12-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: Diabetes; Diabetic Foot; Allograft; Scaffold; Amnion; Chorion; Wound Healing; Advanced Wound Care; Comparative Effectiveness; Lower Extremity Ulcer; Time to heal; Treatment; Diabetes Complication; Skin Ulcer; Neuropathy; Peripheral artery disease; Ischemia; Wagner Grade
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Leg Ulcer; Diabetes Complications; Skin Ulcer; Peripheral Arterial Disease; Ischemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study will be a multicenter, prospective, randomized design in which one treatment group will be compared to one control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FoundationDRS Solo (Experimental): FoundationDRS Solo is a porous, degradable composite scaffold composed of chitosan and chondroitin sulfate
  Interventions: Other: FoundationDRS Solo; Other: Standard of Care
- Standard of Care (Active Comparator): Standard of care (SOC) will include cleansing of the index wound with sterile normal saline solution, followed by sharp debridement to remove necrotic tissue, application of appropriate dressings and wound off-loading.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: FoundationDRS Solo — FoundationDRS Solo is a porous, degradable composite scaffold composed of chitosan and chondroitin sulfate
  Other Names: Foundation DRS
  Arms: FoundationDRS Solo
Other: Standard of Care — Standard of care (SOC) will include cleansing of the index wound with sterile normal saline solution, followed by sharp debridement to remove necrotic tissue, application of appropriate dressings and wound off-loading

SUMMARY:
The goal of this clinical trial is to learn if using FoundationDRS Solo improves healing of chronic, non-healing foot ulcers in diabetic patients.

The main question that this study aims to answer is:

Does FoundationDRS Solo, when used in conjunction with standard of care wound management techniques, result in a higher percentage of target ulcers achieving complete closure (i.e. healing) as compared to ulcers being treated with standard of care alone after 12 weeks of treatment.

One ulcer on each participant's foot will receive weekly applications of 1) FoundationDRS Solo and standard of care wound management or 2) standard of care wound management alone. Pictures of the ulcer and measurements of its size will be measured every week to track its healing progress over a total treatment period of 12 weeks. Additionally, the participants will be asked to fill out a questionnaire about the wound impacts their life and their quality of life.

DETAILED DESCRIPTION:
Patients with diabetes often develop ulcers on their lower extremities. While some ulcers can be managed using standard of care wound management techniques including debridement, moist dressings, infection control and off-loading, many develop into chronic, non-healing wounds. Chronic non-healing wounds can lead to higher risk of infection, amputation and decreased quality of life.

Advanced wound therapies aim to promote rapid and complete healing of chronic wounds. Examples of an advanced wound therapies include scaffolds that contain and / or mimic the structure and function of the natural extracellular matrix of tissue. Several biomimetic scaffolds have been cleared for the management of a variety of wounds (including DFU's) by the US FDA.

The focus of this clinical trial is to determine the clinical utility of treating diabetic foot ulcers with weekly applications of FoundationDRS Solo in addition to standard of care wound management techniques compared to applying standard of care wound management only.

It is hypothesized that the addition of FoundationDRS Solo to standard of care treatment will result in a higher percentage of ulcers achieving complete closure (i.e. healing) compared to ulcer being treated with standard of care alone after 12 weeks of treatment.

To test this hypothesis the study will consist of patients who will undergo standard of care for 4-weeks prior to entering a 12-week treatment phase. During the 4-week standard of care phase, patients meeting inclusion criteria (including confirmation that ulcer does not reduce in area by more than 45%) will be randomized into the treatment groups. During the 12-week treatment phase, index wounds will be treated weekly with FoundationDRS Solo and standard of care or standard of care alone.

Evaluation of data (outcome measures) associated with the trial will include intent to treat and per protocol analyses which will be performed by at least one blinded statistician and investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20.0 cm2 measured post debridement.
4. The target ulcer must have been present for a minimum of 4 weeks and is unresponsive to standard wound care.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. 1. The target ulcer has been present for more than 52 weeks.
2. The ulcer includes exposed tendon or bone.
3. The potential subject is known to have a life expectancy of < 6 months.
4. The potential subject's target ulcer is not secondary to diabetes.
5. The target ulcer is infected or has cellulitis in the surrounding skin.
6. There is evidence of osteomyelitis complicating the target ulcer.
7. The potential subject has an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
8. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
9. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
10. The potential subject has a previous partial amputation on the affected foot that resulted in a deformity impeding proper offloading of the target ulcer.
11. The surface area of the potential subject's target ulcer has reduced in size by more than 45% in the 4 weeks prior to Treatment Visit 1 ("historical" run-in period*) OR the surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit AND the surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV1) to the TV-1 visit.
12. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
13. The potential subject has an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer.
14. The potential subject is pregnant or considering becoming pregnant within the next 6 months.
15. The potential subject has end stage renal disease requiring dialysis.
16. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
17. The potential subject has, in the opinion of the investigator, a medical or psychological condition that may interfere with study assessments.
18. The potential Subject is treated with hyperbaric oxygen therapy or cellular, acellular and matrix-like products (CAMPS) in the 30 days prior to the initial screening visit.
19. A subject is excluded if they are malnourished: a score of less than 17 on the Mini Nutritional Assessment (MNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complete Wound Closure | 12-weeks following study screening phase
  The percentage of wounds completely healed. Complete healing will be defined as 100% epithelialization without drainage and need for dressing or wound size ≤ 0.1cm^2 as determined by the site investigator and validated by a blinded review board.

SECONDARY OUTCOMES:
Time to wound closure | 12-weeks following study screening phase
  Time to wound closure over 12 weeks will be determined via a Kaplan-Meier analysis
Percent reduction in wound area | 12-weeks following study screening phase
  Percent reduction of wound area [(Ai-Axw]) / Ai] x100, where Ai is the area of the index wound at randomization, Axw is the wound area at weekly intervals.
Adverse Events | 12-weeks following study screening phase
  A symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries will be regarded as adverse events. Abnormal results of laboratory or diagnostic procedures are considered to be adverse events if the abnormality:
  Leads to study withdrawal. Is associated with a serious adverse event. Is associated with clinical signs or symptoms. Leads to additional treatment or to further diagnostic tests. Is considered by the Investigator to be of clinical significance
Forgotten Wound Score | 12-weeks following study screening phase
  The forgotten wound score is on a range from 0 to 100, with the higher score indicating a high degree of "forgetting" the wound.
Wound Quality of life (Wound-QoL) questionnaire | 12-weeks following study screening phase
  Average scores will range from 0 (lowest score) to 4 (highest score), with a higher score indicating that the wound effected the subject's quality of life more severely.

OTHER OUTCOMES:
Proportion of ulcers that completely heal in patients 65 years or older | 12-weeks following study screening phase
  Proportion of ulcers that completely heal in patients 65 years or older for CAMP plus SOC versus SOC alone

IPD SHARING:
Plan to Share IPD: No